CLINICAL TRIAL: NCT04431297
Title: The Impact of Virtual Mindfulness Education Sessions on Staff Perceived Stress During COVID-19
Brief Title: Virtual Mindfulness Rounds in the Time of COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jeffrey Zahn, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 20-1022
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Chronic Stress
Keywords: Stress mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Care Workers (Other): Voluntary participation in the virtual presentations
  Interventions: Other: Mindfulness Rounds

INTERVENTIONS:
Other: Mindfulness Rounds — Virtually delivered mindfulness education sessions of 15-30 minutes, two times/week, for four weeks

SUMMARY:
Mindfulness education will be provided via a virtual platform to see if staff stress can be decreased during this time of pandemic.

DETAILED DESCRIPTION:
Healthcare workers have been front and center in battling the COVID crisis. This is a situation the researchers could never have envisioned before it happened. Of course, this has triggered an inordinate amount of stress. Research shows that chronic stress leaves one imbalanced and one's health and happiness to suffer. Research has also demonstrated that how one thinks about stress determines how the body responds to it. Simple mindfulness practices provide healthier ways to deal with stress. In this study, the researchers will introduce modified mindfulness practices that can be practiced in the healthcare setting or at home. All of the practices are based on mindfulness principles. Mindfulness refers to a state of being present in the moment, on purpose, and without judgment. "Mindfulness Based Stress Reduction" is an 8 week, 2 hours/week curriculum that has shown results for over 40 years. All the practices in this study are adapted from that protocol.

The intervention includes several mindfulness practices including an awareness of breath focus instruction, breath-and-body coordination and awareness instruction, and instruction in identifying times to practice these exercises. The intervention will be delivered virtually 2-day/week, twice/day, for four weeks.

Effectiveness will be measured by the voluntary, anonymous submission of a Perceived Stress Scale, a validated survey tool to determine an individual's perceived stress level.

Participants will be healthcare workers and hospital staff in the Mount Sinai Hospital system.

ELIGIBILITY:
Inclusion Criteria:

* Mount Sinai Hospital employee

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale | baseline and Week 6
  Participants will file a 10 question validated survey tool call the Perceived Stress Scale (PSS) before and after the 4-week virtual educational intervention. Total scale range from 0 to 40, higher score indicates more perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zahn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States